CLINICAL TRIAL: NCT07295197
Title: Analysis of Oro-Dental Manifestations for the Screening of Eating Disorders.
Brief Title: Oral Indicators for ED Screening
Acronym: OHEDS
Status: Recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Marco Montevecchi, Researcher, University of Bologna
Other Study IDs: OHEDS
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Eating Disorders; Oral Health; Eating Disorders Symptoms
Keywords: Eating disorders; Oral health; Dental erosion; Oro-dental manifestations; Disordered eating; Screening tool; SCOFF questionnaire; ESP questionnaire; DEQ questionnaire; OHEDs Checklist; OHEDs
MeSH Terms: conditions — Feeding and Eating Disorders; Tooth Erosion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: This is an observational study. No interventions are administered and all assessments are part of routine clinical care.

SUMMARY:
The main objective of this research project is to explore the capability of a standardized, evidence-based study tool (the OHEDs Checklist) in the early identification of oro-dental manifestations potentially indicative of an eating disorder.

The secondary objective is to evaluate the sensitivity and specificity of the OHEDs Checklist in comparison with validated screening instruments for eating disorders, namely the ESP, SCOFF and DEQ questionnaires.

DETAILED DESCRIPTION:
The OHEDS (Oral Health Eating Disorders Screening) study aims to investigate whether specific oro-dental manifestations can be used as early indicators of eating disorders. The project arises from increasing scientific evidence linking various clinical oral signs to disordered eating behaviors, including dental erosion, mucosal alterations, dentin hypersensitivity, changes in salivary flow, and dysfunctional oral hygiene habits. Despite these associations, no structured clinical tool currently exists to interpret such signs as potential early warning indicators.

The OHEDs Checklist was developed from a systematic review of the literature, assigning weighted scores to clinical items based on the consistency and robustness of the available evidence. This study seeks to evaluate the discriminative ability of the Checklist's total score by comparing it with validated screening instruments (SCOFF, ESP, DEQ), with the objective of identifying an optimal cutoff for clinical suspicion.

The study is observational, cross-sectional, and multicentric at a national level. All assessments are performed during routine dental visits already scheduled as part of standard clinical practice, without introducing any experimental interventions. After providing informed consent, participants undergo an intraoral clinical examination conducted by trained clinicians, during which the OHEDs Checklist is completed. Participants also complete validated questionnaires assessing disordered eating behaviors. Demographic, behavioral, and general clinical information is collected according to standard anamnesis procedures.

All data are recorded in pseudonymized form within an electronic Case Report Form (CRF) using the REDCap platform (University of Bologna).

The planned sample size is 461 participants. The first dataset (n = 307) provides adequate precision for estimating the expected prevalence of individuals at risk, while a second independent dataset (n = 154) is used for external validation of the identified cutoff.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Presence of at least 20 permanent teeth (third molars excluded)
* Both males and females are eligible
* Ability to provide written informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Use of systemic antibiotics within the previous month
* Active orthodontic treatment
* Presence of systemic diseases that may affect oral conditions, including: diabetes, ulcerative colitis, Crohn's disease, Sjögren's syndrome, HIV infection, hematologic diseases, neoplasms
* Mental disorders or neuromotor deficits that may interfere with the oro-dental clinical signs evaluated by the OHEDs Checklist
* Use of xerogenic medications or drugs that may alter salivary flow or oral/perioral mucosal conditions, including: antihypertensives, beta-blockers, non-steroidal anti-inflammatory drugs (NSAIDs), antiparkinson medications, anxiolytics, antidepressants, neuroleptics

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Consecutively, all subjects aged 18 to 40 years presenting for routine dental care at the participating centers and meeting the inclusion criteria were enrolled. Eligible participants were required to present at least 20 permanent teeth and provide written informed consent. Subjects with systemic diseases, ongoing orthodontic treatment, recent antibiotic use, pregnancy or breastfeeding, or taking xerogenic or mucosa-altering medications were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 461 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Prevalence of participants classified as "at risk" according to the OHEDs Checklist | Baseline (single assessment during routine dental visit)
  Proportion of participants who receive a score indicating possible risk for eating disorders on the OHEDs Checklist during the single study visit. This outcome shows how many individuals in the sample are classified as "at risk" based on their Checklist score.

SECONDARY OUTCOMES:
Sensitivity, specificity, PPV, NPV and ICC of the OHEDs Checklist | Baseline (single assessment)
  To evaluate the diagnostic performance of the OHEDs Checklist by assessing its sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and intraclass correlation coefficient (ICC) in comparison with validated screening tools for eating disorders (SCOFF and ESP).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontoiatrica - Reparto di Igiene Dentale, Università di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized and aggregated data will be made available upon reasonable request once the study findings have been published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available when the research will be published
Access Criteria: On request to the main investigator

REFERENCES:
- [Result] Valeriani L, Frigerio F, Piciocchi C, Piana G, Montevecchi M, Donini LM, Mocini E. Oro-dental manifestations of eating disorders: a systematic review. J Eat Disord. 2024 Jun 24;12(1):87. doi: 10.1186/s40337-024-01050-8. PMID 38915100
- See also: Italian National Platform for Eating Disorders (ISS) — https://piattaformadisturbialimentari.iss.it/